CLINICAL TRIAL: NCT03123237
Title: Quantitative Renal Uptake Using TC99m DMSA in Hypertensive &/or Diabetic Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebat Allah Ahmed Askar, Principle investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DMSA
Record Dates: First submitted 2017-04-15; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (Placebo Comparator): control will be subjected to:
  • Quantitative Tc99m DMSA renal scan using SPECT technique.
  Interventions: Diagnostic Test: DMSA scan
- Diabetic (Active Comparator): diabetic cases will be subjected to:
  • Quantitative Tc99m DMSA renal scan using SPECT technique.
  Interventions: Diagnostic Test: DMSA scan
- Hypertensive (Active Comparator): hypertesive cases will be subjected to:
  • Quantitative Tc99m DMSA renal scan using SPECT technique.
  Interventions: Diagnostic Test: DMSA scan
- Diabetic & Hypertensive (Active Comparator): Diabetic & Hypertensive cases will be subjected to:
  • Quantitative Tc99m DMSA renal scan using SPECT technique.
  Interventions: Diagnostic Test: DMSA scan

INTERVENTIONS:
Diagnostic Test: DMSA scan — We explore the possible role of DMSA to detect renal affection in diabetic &/or hypertensive patients by detecting difference in counts using Tc 99m DMSA in control & diabetic &/or hypertensive patients.

SUMMARY:
the investigators explore the possible role of DMSA to detect renal affection in diabetic &/or hypertensive patients by detecting difference in counts using Tc 99m DMSA in control & diabetic &/or hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with diabetes (type2), weather controlled or not.

  * Patients with essential hypertension.
  * Patients with diabetes & hypertension.
  * Within normal renal function (urea & creatinine).
  * Control cases may be normal individuals (apparently healthy) like donors for renal transplant.

Exclusion Criteria:

* • Patients with abnormal renal function.

  * Patients with diseases known to affect kidney function rather diabetes & hypertension e.g. SLE, heart failure or liver cell failure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Renal Counts | 2-4 hours
  Quantitative Tc99m DMSA renal scan using SPECT technique will be used to measure renal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt